CLINICAL TRIAL: NCT03659084
Title: Multicenter Prospective Observational Study of the Outcome of Patients With Acute Myeloblastic Leukemia (AML) and Myelodysplastic Syndrome (MDS) Receiving Iron Chelation Therapy (Exjade) After Allogeneic Hematopoietic Stem Cell Transplantation (Allo-HSCT)
Brief Title: Study of the Outcome of Patients With Acute Myeloblastic Leukemia and Myelodysplastic Syndrome Receiving Iron Chelation Therapy After Allogeneic Hematopoietic Stem Cell Transplantation
Acronym: GREFFE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 2013.812
Record Dates: First submitted 2018-08-27; First posted 2018-09-06 (Actual); Last update posted 2018-09-06 (Actual); Status verified 2018-09

CONDITIONS: Myeloid Leukemia; Myelodysplastic Syndromes
Keywords: Acute myeloid leukaemia; Myelodysplastic syndrome; Iron Chelation Therapy (Exjade); allogeneic Hematopoietic Stem Cell transplantation (Allo-HSCT)
MeSH Terms: conditions — Leukemia, Myeloid; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — Deferasirox

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: EXJADE — The patient having given his consent, will begin the Exjade at 10 mg / kg per day if the ferritin level reached 1000 ng / ml at 6 months after allograft, for a minimum duration of three months and up to 6 months. The iron parameters will be evaluated at 3, 6, 9, 12, 18 and 24 months after the beginning of the exjade treatment. The evaluation of the disease will be carried out according to the practices of the center. It is recommended to have a washout period of one week between stopping the ciclosporin and the beginning of treatment by exjade.

SUMMARY:
Iron chelation, mostly associated with multiple red blood cell transfusion, is relatively common in patients with hematological malignancies receiving allo-HSCT.

This multicenter prospective observational study is designed to establish the impact of iron chelation on relapse after allo-HSCT in patients with acute myeloid leukemia and myelodysplastic syndrome. The investigators will compare the results obtained in the prospective study to those observed in a historical retrospective cohort of paired patients who did not receive chelation. Given our clinical experience and literature results, the investigators will evaluate the Exjade chelator. Although not demonstrated, the presence of mutations of the HFE gene could play an indirect role on leukemogenesis by promoting overload. It is therefore important to evaluate the status in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* adults older than 18 years old
* Patients with AML or MDS in complete remission receiving CSH transplantation from a related or unrelated donor and after myeloablative or non-myeloablative conditioning.
* Patients with iron overload defined by at least one ferritinemia> 1000 μg / L in the 6th month after CSH allograft
* Creatinine less than 1.5 x ULN; ALAT and ASAT <2 x ULN
* Patients giving their informed consent (prior to performing any study procedure)

Exclusion Criteria:

* Hypersensitivity to the Exjade
* Association with another iron chelator
* Proteinuria> 1g / 24h
* Acute and chronic hepatitis (B and C viruses); HIV
* Extended corrected QT
* History of ocular toxicity related to iron chelation treatment
* Gastrointestinal Abnormal Absorption of Oral Medications
* Pregnancy and lactation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute leukemia (AML) or Myelodysplastic Syndrome (MDS) and iron overload with ferritinemia ≥ 1000 μg / l, 6 months after CSH allograft.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
Impact of iron chelation on relapse-free survival rate | At 2 years
  Relapse-free survival will be defined as the number of days between the date of diagnosis and the date of death and / or relapse (or censored at the end of follow-up).

SECONDARY OUTCOMES:
Comparison of relapse-free survival after allograft of chelated patients to allografted patients not receiving chelation. | At 2-year
  Matching variables will include disease type (AML or MDS), prognostic factors (cytogenetics, molecular biology, age), donor type / matching, and type of conditioning.
Cumulative incidence of GVHD | 3 months, 1 and 2 years
  Acute and chronic GVHD date and maximum grade using international classification
Rate of infection | Through study completion, an average of 4 years
  during the observation period
Hematological toxicity during administration of Exjade | Through study completion, an average of 4 years
  Hemoglobin level; Current average frequency of transfusions
Non-hematological toxicity during administration of Exjade | Through study completion, an average of 4 years
  Ferritinemia
Non-hematological toxicity during administration of Exjade | Through study completion, an average of 4 years
  Transferrin

CONTACTS AND LOCATIONS:
Overall Officials: Mauricette MICHALLET, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Centre Hospitalier Lyon Sud, Pierre-Bénite, France